CLINICAL TRIAL: NCT07013799
Title: Does Warm-Up Duration Matter? Analyzing the Impact of Three Different Warm-Up Durations on Physical Performance in Highly Trained Youth Basketball Athletes.
Brief Title: Analyzing the Impact of Three Warm-Up Durations on Physical Performance in Youth Basketball Athletes.
Acronym: WUD-YBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-96
Record Dates: First submitted 2025-05-29; First posted 2025-06-10 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Jumping Performance; Speed; Agility
Keywords: Basketball; Sports Performance; Warm-up; Speed; Agility; Jumping Performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short protocol - 5 minutes (Experimental): Participants will perform a condensed version of the BasketUp warm-up, completing only one set of each exercise with minimal repetitions. The focus will remain on basketball-specific mobility, strength, agility, and neurocognitive drills, but in a time-efficient format.
  Interventions: Other: BasketUp Warm-up
- Medium protocol - 10 minutes (Experimental): This group will follow a moderate-duration BasketUp routine, with slightly longer repetitions and 1 to 2 sets per exercise. It will maintain a balance between efficiency and training volume across all three warm-up blocks.
  Interventions: Other: BasketUp Warm-up
- Long protocol - 20 minutes (Experimental): Participants will complete the full-length BasketUp program, including longer repetitions and 2 to 3 sets of each exercise. This version will provide the most comprehensive preparation, emphasizing progressive intensity and volume in mobility, strength, agility, and cognitive components.
  Interventions: Other: BasketUp Warm-up

INTERVENTIONS:
Other: BasketUp Warm-up — BasketUp is a basketball-specific warm-up program designed to meet the sport's physical and physiological demands. Based on the FIFA 11+ structure, it includes three blocks: mobility, strength and plyometrics, and agility with neurocognitive exercises. The program progresses weekly and can be adapted in duration and volume to fit different training needs.

SUMMARY:
This study will explore how different warm-up durations (5, 10, and 20 minutes) affect performance in youth basketball players. Using a basketball-specific routine, it will measure changes in jumping, sprinting, and agility. The goal is to find out which warm-up length best prepares young athletes for high-intensity play.

DETAILED DESCRIPTION:
This study aims to examine the effects of different warm-up durations (5, 10, and 20 minutes) on physical performance in highly trained youth basketball players aged 12-16. Using a standardized basketball-specific warm-up structure (BasketUp), the study will assess how each duration influences key performance outcomes such as vertical jump, agility, and sprint speed. The goal is to determine whether a longer or shorter warm-up is more beneficial for optimizing performance in high-intensity team sports like basketball, providing practical guidance for coaches and sports professionals working with young athletes.

ELIGIBILITY:
Inclusion Criteria:

* At least two years of continuous membership in the squad academy.
* Participation in a minimum of 80% of all training sessions.

Exclusion Criteria:

* Any ongoing injury or discomfort reported by the participant that restricts sports participation.
* A history of injuries treated non-surgically within the last three months.
* A history of injuries treated surgically within the past nine months.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Maximum Jump Height in the Countermovement Jump (CMJ) | Baseline and immediately post-intervention
  The countermovement jump (CMJ) is a common test to assess lower-limb explosive power. Athletes start standing with hands on hips and perform a maximal vertical jump by quickly bending and extending their hips and knees. Two types are tested: bilateral (both legs) and unilateral (one leg). Each athlete performs three attempts per type, resting 30 seconds between jumps. The highest jump height (measured in centimeters) in each modality is recorded as the performance. The higher the jump, the better the performance.
Mean Time to Complete the Cone Drill Test | Baseline and immediately post-intervention
  The Cone Drill test measures agility and the ability to change direction quickly, skills important for basketball performance. Athletes complete a circuit with multiple direction changes as fast as possible. The total time to finish the circuit is recorded using timing sensors. A faster time indicates better agility and performance.
Mean Sprint Time Over 14 and 20 Meters | Baseline and immediately post-intervention.
  Sprint capacity is evaluated over two distances: 14 meters, which reflects typical basketball court movement, and 20 meters, commonly used in sports performance testing. Athletes start from a three-point stance and sprint each distance in a straight line. They rest 60 seconds between sprints, and sprint times are recorded using timing sensors at the start and finish lines. Faster times indicate better sprint performance and acceleration.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Domínguez Navarro, Dr, Principal Investigator — University of Valencia
Locations (1):
- University Cardenal Herrera, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No